CLINICAL TRIAL: NCT03900013
Title: Clinical and Radiographic Evaluation of Injectable PRF With Demineralized Freeze-Dried Bone Allograft (DFDBA) Compared to (DFDBA) in Treatment of Intraosseous Defects in Patients With Stage III Periodontitis: A Randomized Clinical Trial
Brief Title: Injectable Platelet Rich Fibrin With Demineralized Freeze-dried Bone Allograft in Treatment of Intraosseous Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mashaal Mohammed Abdullah Mohammed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MASH2019
Record Dates: First submitted 2019-03-31; First posted 2019-04-02 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Intrabony Periodontal Defect
Keywords: Injectable platelet rich fibrin; I-PRF; Demineralized Freeze-Dried Bone Allograft; DFDBA; Stage 3 periodontitis; 3 wall intraosseous defect; 2 wall intraosseous defect
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the type of intervention, only the outcome assessor and the statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injectable Platelet Rich Fibrin (i-PRF) with DFDBA (Experimental): In i-PRF assigned group, 10 cc of blood per intraosseous defect will be collected right after administering the anaesthesia and will be processed according to the technique proposed by Choukroun et al., 2017 (centrifuged at 700 rpm, for 2-3 minutes). The yellow part will be collected using a syringe and added to a cup that contains the bone grafting material.
  The i-PRF consolidated bone graft will placed into the intraosseous defect.
  Interventions: Procedure: Injectable platelet rich fibrin combined with DFDBA
- Demineralized Freeze-Dried Bone Allograft (DFDBA) alone (Active Comparator): After debridement and intraoperative recordings, in the control group, the bone graft material will be placed in the intraosseous defect without overfilling.
  Interventions: Procedure: Demineralized Freeze Dried Bone Allograft

INTERVENTIONS:
Procedure: Injectable platelet rich fibrin combined with DFDBA — The i-PRF will be mixed with bone graft then will be placed into the intraosseous defect
  Arms: Injectable Platelet Rich Fibrin (i-PRF) with DFDBA
Procedure: Demineralized Freeze Dried Bone Allograft — Demineralized Freeze Dried Bone Allograft alone will be placed into the intraosseous defect
  Arms: Demineralized Freeze-Dried Bone Allograft (DFDBA) alone

SUMMARY:
Clinical and radiographic evaluation of injectable platelet rich fibrin (i-PRF) and demineralized freeze-dried bone allograft (DFDBA) compared to demineralized freeze-dried bone allograft (DFDBA) alone in management of intraosseous defects in stage III periodontitis patients.

DETAILED DESCRIPTION:
Intraosseous defects are defined by the apical location of the periodontal pocket to the alveolar crest. In a recent radiographic study employing cone-beam computed tomography, a high prevalence of intraosseous defects 83% has been reported. Treatment of intraosseous defects is clinically challenging, as they often require complex regenerative periodontal therapy. Current regenerative techniques often employed in treatment of intraosseous defects demonstrate variation in improvement of clinical outcomes and degree of periodontal regeneration achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Type III periodontitis patient having at least one tooth with 2-wall, 3-wall, or combined 2- to 3-wall intraosseous defect ≥ 3 mm in depth (assessed by bone sounding, radiographic examination) with clinical attachment level ≥ 5 mm and pocket depth ≥ 6 mm.
2. Defect not extending to a root furcation area
3. Vital teeth
4. Non-smokers.
5. No history of intake of antibiotics or other medications affecting the periodontium in the previous 6 months.
6. No periodontal therapy carried out in the past 6 months.
7. Able to sign an informed consent form.
8. Patients age between 25 and 50 years old.
9. Patients who are cooperative, motivated, and hygiene conscious.
10. Systemically free according to Cornell Medical Index

Exclusion Criteria:

1. Pregnancy or breast feeding
2. The presence of an orthodontic appliance
3. Teeth mobility greater than grade I

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-10-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level gain (CAL) | CAL will be measured at base line, 3, 6, and 9 months postoperative
  CAL will be measured from the cemento-enamel junction to the bottom of the gingival sulcus/periodontal pocket using the University of North Carolina periodontal probe at six sites per tooth.

SECONDARY OUTCOMES:
Probing Depth (PD) | PD will be measured at base line, 3, 6, and 9 months postoperative
  PD will be measured from the gingival margin to the bottom of the gingival sulcus/ periodontal pocket using the University of North Carolina periodontal probe at six sites per tooth.
Radiographic defect fill (IBD) | Radiographic defect fill will be measured at base line, 6, and 9 months postoperative
  The depth of intrabony defect will be measured from the alveolar bone crest to the base of the defect at baseline, six months and after nine months to detect the amount of bone fill Individually customized bite blocks and parallel-angle technique will be used to obtain standardized radiograph. Radiographs will be scanned and the radiographic defect fill depth will be measured by a computer-aided software program
Gingival Recession Depth (RD) | RD will be measured at base line, 3, 6, and 9 months postoperative
  RD will be measured from the cemento-enamel junction to the most apical extension of the gingival margin using the University of North Carolina periodontal probe at six sites per tooth.
Post-surgical patient satisfaction | After 9 months postoperative
  A 3-item questionnaire will be asked to the patients and shall use a 7-points answer scale. These items will be:
  Would you experience the same surgery another time? Would you advice others with the surgery? To what extent are you satisfied with the results? 7 points mean the best
  1 means the worst

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, Professor, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Castro AB, Meschi N, Temmerman A, Pinto N, Lambrechts P, Teughels W, Quirynen M. Regenerative potential of leucocyte- and platelet-rich fibrin. Part A: intra-bony defects, furcation defects and periodontal plastic surgery. A systematic review and meta-analysis. J Clin Periodontol. 2017 Jan;44(1):67-82. doi: 10.1111/jcpe.12643. Epub 2016 Nov 24. PMID 27783851
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Background] Alsousou J, Thompson M, Hulley P, Noble A, Willett K. The biology of platelet-rich plasma and its application in trauma and orthopaedic surgery: a review of the literature. J Bone Joint Surg Br. 2009 Aug;91(8):987-96. doi: 10.1302/0301-620X.91B8.22546. PMID 19651823
- [Background] Bowers GM, Chadroff B, Carnevale R, Mellonig J, Corio R, Emerson J, Stevens M, Romberg E. Histologic evaluation of new attachment apparatus formation in humans. Part III. J Periodontol. 1989 Dec;60(12):683-93. doi: 10.1902/jop.1989.60.12.683. PMID 2614633
- [Background] BRODMAN K, ERDMANN AJ Jr, LORGE I, GERSHENSON CP, WOLFF HG. The Cornell Medical Index-health questionnaire. IV. The recognition of emotional disturbances in a general hospital. J Clin Psychol. 1952 May;8(3):289-93. doi: 10.1002/1097-4679(195207)8:33.0.co;2-b. No abstract available. PMID 12981181
- [Background] Chang YC, Zhao JH. Effects of platelet-rich fibrin on human periodontal ligament fibroblasts and application for periodontal infrabony defects. Aust Dent J. 2011 Dec;56(4):365-71. doi: 10.1111/j.1834-7819.2011.01362.x. Epub 2011 Oct 13. PMID 22126345
- [Background] Chenchev IL, Ivanova VV, Neychev DZ, Cholakova RB. Application of Platelet-Rich Fibrin and Injectable Platelet-Rich Fibrin in Combination of Bone Substitute Material for Alveolar Ridge Augmentation - a Case Report. Folia Med (Plovdiv). 2017 Sep 1;59(3):362-366. doi: 10.1515/folmed-2017-0044. PMID 28976904
- [Background] Del Corso M, Vervelle A, Simonpieri A, Jimbo R, Inchingolo F, Sammartino G, Dohan Ehrenfest DM. Current knowledge and perspectives for the use of platelet-rich plasma (PRP) and platelet-rich fibrin (PRF) in oral and maxillofacial surgery part 1: Periodontal and dentoalveolar surgery. Curr Pharm Biotechnol. 2012 Jun;13(7):1207-30. doi: 10.2174/138920112800624391. PMID 21740371